CLINICAL TRIAL: NCT00542373
Title: Fluorescence & Reflectance Imaging to Detect Oral Neoplasia
Brief Title: Widefield Fluorescence and Reflectance Imaging Systems and Oral Tissue Samples in Monitoring Participants at Risk for Developing Oral Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0802; P30CA016672 (NIH); NCI-2015-01903 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0802 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Erythroplakia; Fanconi Anemia; Lichen Planus; Oral Cavity and Lip Precancerous Condition; Oral Cavity Leukoplakia; Oral Neoplasm; Premalignant Lesion; Tobacco Use Disorder
MeSH Terms: conditions — Erythroplasia; Fanconi Anemia; Lichen Planus; Leukokeratosis, Hereditary Mucosal; Mouth Neoplasms; Tobacco Use Disorder | interventions — Molecular Diagnostic Techniques; Optical Imaging; Spectrometry, Fluorescence

ARMS (1):
- Diagnostic (fluorescent/reflectance imaging, spectroscopy) (Experimental): Participants' oral cavities are inspected by a clinician using a standard white light headlamp. Participants then undergo oral mucosa examination using wide-field reflectance and fluorescence imaging, and/or fluorescence spectroscopy imaging. Standard oral brush biopsies are also performed and examined microscopically. Participants may undergo repeated imaging procedures and biopsy during subsequent follow up visits.
  Interventions: Other: Cytology Specimen Collection Procedure; Procedure: Diagnostic Microscopy; Procedure: Diagnostic Procedure; Procedure: Fluorescence Imaging; Procedure: Fluorescence Spectroscopy

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo oral tissue collection
  Other Names: Cytologic Sampling
Procedure: Diagnostic Microscopy — Mouth tissue examined microscopically for cytologic features
Procedure: Diagnostic Procedure — Undergo standard white light headlamp oral examination
  Other Names: Diagnostic Method; Diagnostic Technique; Diagnostic Test
Procedure: Fluorescence Imaging — Undergo widefield fluorescent and reflectance imaging
Procedure: Fluorescence Spectroscopy — Undergo point fluorescent spectroscopy
  Other Names: Spectroscopy, Fluorescence

SUMMARY:
This clinical trial studies widefield fluorescence and reflectance imaging, fluorescence spectroscopy, and tissue samples in regularly examining (monitoring) participants at risk for developing oral cancer. All tissue and cells are made of tiny particles. Some of these particles give off small amounts of light. This light is called fluorescence. Fluorescent imaging use instruments that shine different wavelengths (colors) of light in the mouth taking fluorescence pictures through a portable head light or by taking fluorescent and reflectance pictures through a dental microscope using a digital camera. Fluorescent spectroscopy uses a small probe placed gently against the lining of the mouth and the tissue is exposed to small amounts of fluorescent light that is then collected with a special camera and a computer to be analyzed. Checking mouth tissue samples under a microscope may also help detect abnormal cells. Diagnostic procedures, such as fluorescence and reflectance imaging, fluorescence spectroscopy imaging, and tissue samples, may help doctors detect pre-cancer or early cancer when it may be easier to treat.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare images of oral mucosa, obtained at various wavelength combinations including 350 nm, 380 nm, 400 nm, and 450 nm excitation, to standard white light images, pathologic analysis of any biopsied tissue when available, and carcinogenic progression.

OUTLINE:

Participants' oral cavities are inspected by a clinician using a standard white light headlamp. Participants then undergo oral mucosa examination using wide-field reflectance and fluorescence imaging, and/or fluorescence spectroscopy imaging. Standard oral brush biopsies are also performed and examined microscopically. Participants may undergo repeated imaging procedures and biopsy during subsequent follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with premalignant lesion, or potentially premalignant lesion, of the oral cavity mucosa (leukoplakia or erythroplakia)
* Patients with a history of head and neck cancer or oral premalignant disease but without any clinical evidence of disease
* Persons with any other condition (such as lichen planus, Fanconi anemia, heavy tobacco use, etc) making them at higher risk for oral cancer development
* Patients with either pre-malignant or a history of oral cancer based on patient history and clinical presentations

Exclusion Criteria:

* Subjects under the age of 18.
* Subjects that are unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2007-08-27 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Lesions diagnosed via wide-field fluorescence imaging | Up to 10 years
  Oral mucosa obtained at various wavelength combinations including 350 nm, 380 nm, 400 nm, and 450 nm excitation will be compared to standard white light images, pathologic analysis of any biopsied tissue when available, and carcinogenic progression. Diagnostic methods will be compared with each other by forming 2x2 tables and computing the chi-square statistics for the McNemar test. Kappa statistic will also be calculated for comparing the chance corrected agreement between various diagnostic methods.
Lesions diagnosed via point spectroscopy system | Up to 10 years
  Oral mucosa obtained at various wavelength combinations including 350 nm, 380 nm, 400 nm, and 450 nm excitation will be compared to standard white light images, pathologic analysis of any biopsied tissue when available, and carcinogenic progression. Diagnostic methods will be compared with each other by forming 2x2 tables and computing the chi-square statistics for the McNemar test. Kappa statistic will also be calculated for comparing the chance corrected agreement between various diagnostic methods.
Lesions diagnosed via non-invasive brush cytology | Up to 10 years
  Oral mucosa obtained at various wavelength combinations including 350 nm, 380 nm, 400 nm, and 450 nm excitation will be compared to standard white light images, pathologic analysis of any biopsied tissue when available, and carcinogenic progression. Diagnostic methods will be compared with each other by forming 2x2 tables and computing the chi-square statistics for the McNemar test. Kappa statistic will also be calculated for comparing the chance corrected agreement between various diagnostic methods.

CONTACTS AND LOCATIONS:
Overall Officials: Ann M Gillenwater, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org